CLINICAL TRIAL: NCT06623162
Title: Selective Bladder-Sparing Trial with Sasanlimab As Maintenance Treatment Based on Clinical Response to Neoadjuvant Treatment in Molecularly Categorized Muscle Invasive Bladder Cancer Patients
Brief Title: Sasanlimab As Maintenance Treatment Based on Clinical Response to Neoadjuvant Treatment in Molecularly Categorized Muscle Invasive Bladder Cancer Patients
Acronym: SASAN-SPARING
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación de investigación HM (Other)
Collaborators: MFAR Clinical Research S.L. (Unknown); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-87884561; EU CT (Registry Identifier: 2024-511358-36-00)
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Mibc; Muscle Invasive Bladder Cancer
Keywords: MIBC; sparing; cystectomy; muscle invasive bladder cancer; gemcitabine; cisplatine
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant (Experimental): 4 cycles of gemcitabine plus cisplatin
  Interventions: Drug: gemcitabine + cisplatine

INTERVENTIONS:
Drug: gemcitabine + cisplatine — 4 cycles

SUMMARY:
Selective Bladder-Sparing Trial with Sasanlimab as Maintenance Treatment Based On Clinical Response To Neoadjuvant Treatment In Molecularly Categorized Muscle Invasive Bladder Cancer Patients

DETAILED DESCRIPTION:
All patients will receive 4 cycles of gemcitabine plus cisplatin followed by clinical restaging (Fig.1). After neoadjuvant chemotherapy, patients will be restaged and patients achieving a clinical response (normal cytology, imaging, and cT0/Ta/T1/Tis) will be eligible to proceed without cystectomy and receive maintenance with sasanlimab 300 mg subcutaneous (two product presentations: a vial and a prefilled syringe) every 4 weeks (Q4W) for up to 12 cycles initiating between 3-6 weeks and followed by surveillance (Fig.1). Treatment may be discontinued in case of progression, unacceptable toxicity, patient withdrawal or death. Patients with persistent non-muscle invasive disease (cTa/T1/Tis) at the first evaluation at 12 weeks of maintenance ( after 3 cycles of sasanlimab), will be recommended to undergo cystectomy.

Non clinically responding patients (≥ T2) after neoadjuvant chemotherapy will undergo cystectomy (Fig.1). Patients may undergo late cystectomy throughout the study period in the case of local relapse, following the investigator criteria or according to the patient's choice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign a written informed consent approved by an IEC for the participation in this trial.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of ≤ 1 within 28 days prior to registration (Appendix 6).
4. Histological evidence of localized muscle-invasive urothelial cancer of the bladder (i.e., pT2-T4 / N0 / M0). Candidate for cystectomy as per treating physician.
5. Absence of metastasis as confirmed by CT or MRI scan of pelvis, abdomen and chest no more than 4 weeks pre-enrolenrment.
6. Patients candidates to receive neoadjuvant therapy with gemcitabine and cisplatin. Note:MVAC treatment will not be allowed.
7. All subjects must have adequate archival tissue identified at screening (i.e., at least 15 unstained slides or paraffin block). Subjects without archival tissue must be discussed with the Sponsor-investigator.
8. Adequate organ and bone marrow function as defined below:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   2. Hemoglobin (HgB) ≥ 9 g/dL.
   3. Platelet count ≥ 100 x 10^9/L.
   4. Creatinine ≤ 1.5 or creatinine clearance ≥ 60 mL/min (Cockcroft-Gault formula).
   5. Bilirubin ≤ 1.5 × upper limit of normal (ULN). Note: subjects with Gilbert Syndrome, who have total bilirubin < 3.0 mg/dL are eligible.
   6. Hepatic enzymes Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 3 x ULN.
9. Female patients must either:

   a. Be of nonchildbearing potential: i. Postmenopausal *(defined as at least 1 year without any menses) prior to screening , or ii. Documented surgically sterile (e.g. hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion).
   * Those who are amenorrheic due to an alternative medical cause are not considered postmenopausal and must follow the criteria for childbearing potential subjects. OR b. If of childbearing potential: i. Agree not to try to become pregnant during the study and for at least 6 months after the final study drug administration, ii. And have a negative urine or serum pregnancy test within 7 days prior to Day 1 (females with false positive results and documented verification of negative pregnancy status are eligible for participation), iii. And if heterosexually active, agree to abstinence (if in line with the usual preferred lifestyle of the patient) or consistently use a condom plus 1 form of highly effective birth control (Appendix 7) per locally accepted standards starting at screening and throughout the study period and for at least 6 months after the final study drug administration.
10. Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
11. Male patients with a partner with childbearing potential, or who is pregnant or breastfeeding must agree to abstinence or use a condom plus 1 form of highly effective birth control throughout the study period and for at least 6 months after the final study drug administration.
12. Male patients must not donate sperm starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
14. Patient agrees not to participate in another interventional study while on treatment in the present study

Exclusion Criteria:

* 1. Prior treatment with systemic chemotherapy or other approved anticancer treatments for muscle-invasive urothelial cancer of the bladder. Note: In case of prior non muscle-invasive bladder cancer NMIBC, Mitomycin or Bacillus Calmette Guerin (BCG) treatment are allowed.

  2. Another malignancy that is progressing or required active treatment , with the exception of those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ).

  3. Active or prior autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Note: Patients with diabetes type I, vitiligo, psoriasis, or hypothyroid or hyperthyroid disease not requiring immunosuppressive treatment are eligible.

  4. Patients that have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 28 days prior to the first dose of trial treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses (which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid).

  5. History of allogeneic organ transplant. 6. Active non-infectious pneumonitis, pulmonary fibrosis, or known history of immune mediated pneumonitis.

  7. Active infection requiring systemic therapy. Patients with active, uncontrolled bacterial, fungal, or viral infection, including HBV, HCV, or known HIV infection.

  8. Live attenuated vaccines within 4 weeks prior to the first dose of sasanlimab and through 30 days following the last dose of sasanlimab are not allowed.

Note: influenza and SARS-CoV-2 vaccines which are inactivated are allowed. 9. Clinically significant cardiovascular diseases, including any of the following:

1. History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) ≤6 months prior to start of study treatment.
2. Congestive heart failure requiring treatment (New York Heart Association Class ≥2).
3. Uncontrolled hypertension, defined as persistent systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg despite optimal therapy.
4. History or presence of clinically significant or uncontrolled sustained cardiac arrhythmias (including uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia).
5. History of thromboembolic or cerebrovascular events ≤3 months prior to the first dose of study treatment, including ischemic attacks, cerebrovascular accidents, hemodynamically significant (ie, massive or sub-massive) deep vein thrombosis or pulmonary emboli. Note: Participants with either deep vein thrombosis or pulmonary emboli that do not result in hemodynamic instability are allowed to enroll as long as they are stable, asymptomatic and on stable anticoagulants for at least 2 weeks. Note: Participants with thromboembolic events related to indwelling catheters or other procedures may be enrolled. 10. Major surgery less than 28 days prior to the first dose of study treatment. 11. Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis.

   12. Known or suspected hypersensitivity to active ingredients or excipients of the study drug.

   13. Pregnant or breastfeeding. 14. Any serious or uncontrolled medical disorder, psychiatric or social condition that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the bladder-intact overall survival at 12 months after the first dose of sasanlimab. Bladder-intact overall survival is defined as the time from initiation of sasanlimab treatment until death or cystectomy | 12 months
  The primary endpoint will be the bladder-intact overall survival rate at 12 months after the first dose of sasanlimab. Bladder-intact overall survival is defined as the time from initiation of sasanlimab treatment until death or cystectomy. The primary endpoint will be the percentage of patients who are alive and with no cystectomy at 12 months after the first dose of sasanlimab.

CONTACTS AND LOCATIONS:
Locations (1):
- Hm Sanchinarro, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Background] Bruck K, Meijer RP, Boormans JL, Kiemeney LA, Witjes JA, van Hoogstraten LMC, van der Heijden MS, Donders AR, Franckena M, Uyl de Groot CA, Leliveld AM, Aben KKH, Hulshof MCCM. Disease-Free Survival of Patients With Muscle-Invasive Bladder Cancer Treated With Radical Cystectomy Versus Bladder-Preserving Therapy: A Nationwide Study. Int J Radiat Oncol Biol Phys. 2024 Jan 1;118(1):41-49. doi: 10.1016/j.ijrobp.2023.07.027. Epub 2023 Jul 28. PMID 37517601
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Brahmer JR, Abu-Sbeih H, Ascierto PA, Brufsky J, Cappelli LC, Cortazar FB, Gerber DE, Hamad L, Hansen E, Johnson DB, Lacouture ME, Masters GA, Naidoo J, Nanni M, Perales MA, Puzanov I, Santomasso BD, Shanbhag SP, Sharma R, Skondra D, Sosman JA, Turner M, Ernstoff MS. Society for Immunotherapy of Cancer (SITC) clinical practice guideline on immune checkpoint inhibitor-related adverse events. J Immunother Cancer. 2021 Jun;9(6):e002435. doi: 10.1136/jitc-2021-002435. PMID 34172516
- [Background] Bellmunt J, Hussain M, Gschwend JE, Albers P, Oudard S, Castellano D, Daneshmand S, Nishiyama H, Majchrowicz M, Degaonkar V, Shi Y, Mariathasan S, Grivas P, Drakaki A, O'Donnell PH, Rosenberg JE, Geynisman DM, Petrylak DP, Hoffman-Censits J, Bedke J, Kalebasty AR, Zakharia Y, van der Heijden MS, Sternberg CN, Davarpanah NN, Powles T; IMvigor010 Study Group. Adjuvant atezolizumab versus observation in muscle-invasive urothelial carcinoma (IMvigor010): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Apr;22(4):525-537. doi: 10.1016/S1470-2045(21)00004-8. Epub 2021 Mar 12. PMID 33721560
- [Background] Balar et al. 2021 Balar AV, Milowsky MI, O'Donnell PH, et al. Pembrolizumab (pembro) in combination with gemcitabine (Gem) and concurrent hypofractionated radiation therapy (RT) as bladder sparing treatment for muscle-invasive urothelial cancer of the bladder (MIBC): A multicenter phase 2 trial. J. Clin. Oncol. 2021;39:4504.
- [Background] Bajorin DF, Witjes JA, Gschwend JE, Schenker M, Valderrama BP, Tomita Y, Bamias A, Lebret T, Shariat SF, Park SH, Ye D, Agerbaek M, Enting D, McDermott R, Gajate P, Peer A, Milowsky MI, Nosov A, Neif Antonio J Jr, Tupikowski K, Toms L, Fischer BS, Qureshi A, Collette S, Unsal-Kacmaz K, Broughton E, Zardavas D, Koon HB, Galsky MD. Adjuvant Nivolumab versus Placebo in Muscle-Invasive Urothelial Carcinoma. N Engl J Med. 2021 Jun 3;384(22):2102-2114. doi: 10.1056/NEJMoa2034442. PMID 34077643
- [Background] Al-Khami AA, Youssef S, Abdiche Y, Nguyen H, Chou J, Kimberlin CR, Chin SM, Kamperschroer C, Jessen B, Kern B, Budimir N, Dillon CP, Xu A, Clark JD, Chou J, Kraynov E, Rajpal A, Lin JC, Salek-Ardakani S. Pharmacologic Properties and Preclinical Activity of Sasanlimab, A High-affinity Engineered Anti-Human PD-1 Antibody. Mol Cancer Ther. 2020 Oct;19(10):2105-2116. doi: 10.1158/1535-7163.MCT-20-0093. Epub 2020 Aug 26. PMID 32847983
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524